CLINICAL TRIAL: NCT03408561
Title: The Use of Social Media Listening for Targeted Recruitment of Twitter Users in LA County in Cancer Trials Compared to Historic Recruitment Data: A Mixed-Methods Study
Brief Title: Social Media Listening in Improving Clinical Trial Recruitment in Patients With Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0S-17-7; NCI-2017-02145 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-17-7 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Breast Carcinoma; Colon Carcinoma; Kidney Carcinoma; Lymphoma; Non-Small Cell Lung Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Carcinoma, Renal Cell; Lymphoma; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health Services Research (message via Twitter) (Experimental): Patients who mention specific cancer disease keywords and/or hashtags are identified and receive a message via Twitter. Patients are then contacted for recruitment into a clinical trial.
  Interventions: Other: Internet-Based Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Receive message via Twitter
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well social media listening works in improving clinical trial recruitment in patients with cancer. Social media listening and recruitment on Twitter may enhance enrollment for cancer-related clinical trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the feasibility (acceptance among University of Southern California [USC] Norris study team members and Twitter users in Los Angeles [LA] county) of targeted social media listening (SML) via Twitter as a tool for enhancing recruitment to cancer trials.

II. Gain preliminary data on the impact (i.e., numbers recruited versus projected accrual compared to historic recruitment) of targeted social media listening (SML) as a tool for enhancing recruitment to cancer trials among Twitter users in LA county.

III. Estimate the effect size of the number of people enrolled associated with the use of targeted social media listening (SML) via Twitter as a tool for enhancing recruitment to cancer trials.

OUTLINE:

Patients who mention specific cancer disease keywords and/or hashtags are identified and receive a message via Twitter. Patients are then contacted for recruitment into a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* TRIAL INCLUSION:
* Focus on one of the following disease categories: non-small cell lung cancer, colon cancer, breast cancer, prostate cancer, kidney cancer, lymphoma
* Be a phase 1 trial in expansion, phase 2, or 3
* Be interventional trials
* Recruit in English
* Be Institutional Review Board (IRB)-approved and open to accrual at USC Norris
* Recruit for at least 9 months at the point of enrollment
* Set monthly accrual target >= 1/ and annual accrual target >= 12
* PATIENT INCLUSION:
* Will include all prospective trial participants in this study that come from Twitter in response of our SM recruitment interventions, provided they meet the specific trial's eligibility criteria

Exclusion Criteria:

* TRIAL EXCLUSION:
* Phase 1 trials in dose escalation
* PATIENT EXCLUSION:
* Persons who do not meet the eligibility criteria of any of the trials open to accrual will be excluded from participation, and persons who may be eligible (e.g., disease/histology, stage, prior treatment) but do not meet additional trial-specific requirements such as insurance or allergy to drug)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
User acceptance and satisfaction with social media (SM) as a recruitment method | Up to 14 months
  A questionnaire will be used assess the acceptance of and satisfaction with SM recruitment method among University of Southern California (USC) Norris study team members and Twitter users in Los Angeles (LA) county.
Accrual rate | Up to 14 months
  To be determined by comparing monthly actual versus (vs.) projected rate of recruitment for the trial disease groups (i.e., non-small cell lung cancer, colon cancer, breast cancer, prostate cancer, kidney cancer, lymphoma) using generalized estimating equations, accounting for intra-disease random effects and trends across the 12 months (9 months exposure per trial). These results will then be put into context of the historic recruitment for these diseases at the center.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Buchanan, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Reuter K, Angyan P, Le N, Buchanan TA. Using Patient-Generated Health Data From Twitter to Identify, Engage, and Recruit Cancer Survivors in Clinical Trials in Los Angeles County: Evaluation of a Feasibility Study. JMIR Form Res. 2021 Nov 26;5(11):e29958. doi: 10.2196/29958. PMID 34842538
- [Derived] Reuter K, Angyan P, Le N, MacLennan A, Cole S, Bluthenthal RN, Lane CJ, El-Khoueiry AB, Buchanan TA. Monitoring Twitter Conversations for Targeted Recruitment in Cancer Trials in Los Angeles County: Protocol for a Mixed-Methods Pilot Study. JMIR Res Protoc. 2018 Sep 25;7(9):e177. doi: 10.2196/resprot.9762. PMID 30274964